CLINICAL TRIAL: NCT05672316
Title: A Phase I/II Trial of Botensilimab, Balstilimab and Regorafenib (BBR) in Patients With Microsatellite Stable (MSS) Metastatic Colorectal Cancer Who Progressed on Prior Chemotherapy
Brief Title: Botensilimab, Balstilimab and Regorafenib for the Treatment of Patients With Microsatellite Stable Metastatic Colorectal Cancer Who Have Progressed on Prior Chemotherapy
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22351; NCI-2022-10069 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22351 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Advanced Colorectal Adenocarcinoma; Advanced Microsatellite Stable Colorectal Carcinoma; Metastatic Colorectal Adenocarcinoma; Metastatic Microsatellite Stable Colorectal Carcinoma; Stage III Colorectal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — balstilimab; Specimen Handling; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (botensilimab, balstilimab and regorafenib) (Experimental): Patients receive botensilimab IV, balstilimab IV, and regorafenib PO on study. Patients also undergo CT and collection of blood throughout the study.
  Interventions: Biological: Balstilimab; Procedure: Biospecimen Collection; Biological: Botensilimab; Procedure: Computed Tomography; Drug: Regorafenib

INTERVENTIONS:
Biological: Balstilimab — Given IV
  Other Names: AGEN 2034; AGEN-2034; AGEN2034
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Botensilimab — Given IV
  Other Names: AGEN 1181; AGEN-1181; AGEN1181; Anti-CTLA-4 Monoclonal Antibody AGEN1181
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Regorafenib — Given PO
  Other Names: BAY 73-4506; Regorafenib Anhydrous

SUMMARY:
This phase I/II trial tests how well botensilimab, balstilimab, and regorafenib works in treating patients with microsatellite stable colorectal cancer that has spread from where it first started (primary site) to other places in the body (metastatic) or that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) and who have progressed on prior chemotherapy. Immunotherapy with monoclonal antibodies, such as botensilimab and balstilimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Regorafenib binds to and inhibits growth factor receptors, which may inhibit the growth of new blood vessels that tumors need to grow. Giving botensilimab, balstilimab, and regorafenib in combination may work better in treating patients with metastatic colorectal cancer than giving these drugs alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify the recommended phase 2 dose (RP2D) of botensilimab, balstilimab, and regorafenib (BBR) in patients with chemotherapy-resistant microsatellite stable (MSS) metastatic colorectal cancer (MSS mCRC). (Phase I) II. To estimate the overall response rate (ORR) of botensilimab, balstilimab, and regorafenib in patients with chemotherapy-resistant MSS mCRC, with and without liver metastatic disease. (Phase II)

SECONDARY OBJECTIVES:

I. Describe the safety of botensilimab, balstilimab, and regorafenib at all evaluable dose levels. (Phase I) II. Describe the efficacy of BBR in terms of ORR, progression free survival (PFS) and overall survival (OS). (Phase I) III. To evaluate the safety/feasibility of botensilimab, balstilimab, and regorafenib through the assessment of adverse events. (Phase II) IV. Estimate the PFS, OS and duration of response (DOR). (Phase II)

CORRELATIVE OBJECTIVES:

I. Evaluate potential circulating biomarkers of response, resistance, activity, and toxicity. (Phase I/II) II. Correlate baseline molecular biomarkers (RAS, BRAF, TMB, and PD-L1 if available), with overall outcome. (Phase I/II)

OUTLINE: This is a phase I, dose-escalation study of botensilimab followed by a phase II study.

Patients receive botensilimab intravenously (IV), balstilimab IV, and regorafenib orally (PO) on study. Patients also undergo computed tomography (CT) and collection of blood throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines
* Age: >= 18 years
* Eastern Cooperative Oncology Group (ECOG) =< 1
* Life expectancy >= 3 months
* Able to swallow and absorb oral tablets
* Histological or cytological confirmed advanced, metastatic, or progressive proficient mismatch repair (pMMR)/MSS adenocarcinoma of colon or rectum

  * Microsatellite status should be performed per local standard of practice (e.g., immunohistochemistry [IHC] and/or polymerase chain reaction [PCR], or next-generation sequencing). Only participants with pMMR/MSS mCRC are eligible
* Patients should have measurable metastatic disease as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 guidelines
* Known extended RAS and BRAF status as per local standard of practice. TMB and PD-L1 status will be collected when available but not mandated for enrollment
* Patients must have progressed following exposure to all of the following agents:

  * Fluoropyrimidines (capecitabine or 5-FU)
  * Irinotecan
  * Oxaliplatin
  * Anti-EGFR therapy if RAS and BRAF wild type with left colon primary
* Patients must have evidence of progression on or after the last treatment received and within 6 months prior to study enrollment

  * Patients who were intolerant to prior systemic chemotherapy regimens are eligible if there is documented evidence of clinically significant intolerance despite adequate supportive measures
  * Adjuvant/neoadjuvant chemotherapy can be considered as one line of chemotherapy for advanced/metastatic disease if the participant had disease recurrence within 6 months of completion
* For patients with liver metastatic disease, patients must have no more than 5 hepatic metastases at the time of enrollment
* Patients without liver metastatic disease should be either with no history of liver metastatic disease or with history of resected or ablated liver metastases without evidence of disease recurrence in the liver for at least 6 months before enrollment
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (to be performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)
* Aspartate aminotransferase (AST) =< 2.5 x ULN, unless presence of liver metastases for which =< 5 x ULN is allowed (to be performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)
* Alanine aminotransferase (ALT) =< 2.5 x ULN, unless presence of liver metastases for which =< 5 x ULN is allowed (to be performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)
* Serum creatinine =< 1.5 x ULN or creatinine clearance >= 40 mL/min (measured or calculated using the Cockcroft-Gault formula) (to be performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)
* White blood cell (WBC) >= 2000/ul (to be performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)
* Hemoglobin >= 9 g/dl (to be performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)
* Absolute neutrophil count (ANC) >= 1500/ul (to be performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)
* Platelets >= 75,000/mm^3 (to be performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)
* Albumin >= 3.0 g/dl (to be performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required (to be performed within 7 days prior to day 1 of protocol therapy unless otherwise stated)
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from sexual activity for the course of the study through at least 120 days after the last dose of protocol therapy

  * Females of non-childbearing potential defined as:

    * >= 50 years of age and has not had menses for greater than 1 year
    * Amenorrheic for >= 2 years without a hysterectomy and bilateral oophorectomy and a follicle stimulating hormone value in the postmenopausal range upon pre-study (screening) evaluation
    * Status is post-hysterectomy, bilateral oophorectomy, or tubal ligation

Exclusion Criteria:

* Prior immunotherapy with PD-1 or PD-L1 or CTLA-4 targeting agents
* Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) within 14 days or another immunosuppressive medication within 30 days of the first dose of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses =< 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* Prior allogeneic organ transplantation
* Surgical intervention within 4 weeks prior to study treatment, except for minor procedures such as port placement
* Prior allergic reaction or hypersensitivity to any of the study drug components
* Active autoimmune disease or history of autoimmune disease that required systemic treatment within 2 years before starting treatment, i.e., with use of disease-modifying agents or immunosuppressive drugs
* Uncontrolled hypertension, defined as systolic blood pressure (SBP) > 150, diastolic blood pressure (DBP) > 90
* History of acute thrombotic venous events in the last 30 days before enrollment. If within 30 days, the patient should be on anticoagulants and without symptoms
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 12 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class >= III), or serious uncontrolled cardiac arrhythmia requiring medication
* Obstructive bowel symptoms related to unresected primary or carcinomatosis
* Any persistent toxicities (Common Terminology Criteria for Adverse Events [CTCAE] grade >= 2) from prior cancer therapy, excluding endocrinopathies stable on medication, stable neuropathy that is grade 1 or less, and alopecia
* Non-healing wounds
* Symptomatic active bleeding
* Active brain metastases or leptomeningeal metastases with the following exceptions:

  * Treated brain metastases require a) surgical resection, or b) stereotactic radiosurgery. These patients must be off steroids >= 10 days prior to randomization for the purpose of managing their brain metastases. Repeat brain imaging following surgical resection or stereotactic radiosurgery at least 4 weeks from treatment should document lack of progression
* Concurrent non-colorectal second malignancy (present during screening) requiring treatment or history of a non-colorectal second primary metastatic malignancy within 2 years prior to the first dose of study treatment. Patients with history of prior early-stage basal/squamous cell skin cancer, low-risk prostate cancer eligible for active surveillance or noninvasive or in situ cancers who have undergone definitive treatment at any time are also eligible
* Any evidence of current interstitial lung disease (ILD) or pneumonitis or a prior history of ILD or non-infectious pneumonitis requiring high-dose glucocorticoids
* Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* History or current evidence of any condition, co-morbidity, therapy, any active infections, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Known previous SARS-CoV-2 infection within 10 days for mild or asymptomatic infections or 20 days for severe/critical illness prior to cycle 1 day 1 (C1D1)
* Uncontrolled infection with human immunodeficiency virus (HIV). Patients on stable highly active antiretroviral therapy (HAART) with undetectable viral load and normal CD4 counts for at least 6 months prior to study entry are eligible. Serological testing for HIV at screening is not required
* Known to be positive for hepatitis B virus (HBV) surface antigen, or any other positive test for HBV indicating acute or chronic infection. Patients who are receiving or who have received anti-HBV therapy and have undetectable HBV deoxyribonucleic acid (DNA) for at least 6 months prior to study entry are eligible. Serological testing for HBV at screening is not required
* Known active hepatitis C virus (HCV) as determined by positive serology and confirmed by polymerase chain reaction (PCR). Patients on or who have received antiretroviral therapy are eligible provided they are virus-free by PCR for at least 6 months prior to study entry. Serological testing for HCV at screening is not required
* Dependence on total parenteral nutrition or intravenous hydration
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose of botensilimab, balstilimab, and regorafenib (Phase I) | Cycle 1 (6 weeks)
  Will conduct a Simon 2-stage optimal design study.
Incidence of dose limiting toxicities (DLT) (Phase I) | Cycle 1 (6 weeks)
  Graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.
Overall response rate (ORR) (Phase II) | Up to 2 years
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1.

SECONDARY OUTCOMES:
Incidence of DLTs (Phase I) | Up to 2 years
  Graded according to the NCI CTCAE v.5.0.
ORR (Phase I) | Up to 2 years
  Assessed by RECIST 1.1.
Progression-free survival (PFS) (Phase I) | Time to disease progression/ relapse or death as a result of any cause, assessed up to 2 years
Overall survival (OS) (Phase I) | Time to death as a result of any cause, assessed up to 2 years
PFS (Phase II) | Time to disease progression or death as a result of any cause, assessed up to 2 years
OS (Phase II) | Time to death as a result of any cause, assessed up to 2 years
Duration of response (Phase II) | Time to progression or death, starting at the time when a response is experienced, assessed up to 2 years
Incidence of toxicity (Phase II) | Up to 2 years
  Graded according to the NCI CTCAE v.5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Marwan G Fakih, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States